CLINICAL TRIAL: NCT03819634
Title: Longevity of Multi-Slitted Catheter, the Convatec Inset II With Lantern Technology
Brief Title: Longevity of Multi-Slitted Catheter With Lantern Technology
Acronym: Lantern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Principal Investigator, Bruce Buckingham, Professor of Pediatric Endocrinology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #45812
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Insulin Dependent Diabetes Mellitus 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: To determine length of infusion set wear for up to a maximum of 10 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Lantern infusion set (Experimental): Multi-slitted lantern infusion set
  Interventions: Device: Inset II with Lantern Technology

INTERVENTIONS:
Device: Inset II with Lantern Technology — Each participant will insert the Inset II with Lantern technology and wear it for 10 days or until set failure and data will be collected on the cause of set failure. The infusion set will be used with their usual insulin pump.

SUMMARY:
To determine time to set failure when the Convatec Inset II with Lantern technology (Convatec Lantern) infusion set with multi-slitted catheter is worn for up to 10 days

DETAILED DESCRIPTION:
This is a pilot study to obtain preliminary data to determine the time to set failure when the Lantern infusion set is worn for up to 10 days. The study is not intended for registration purposes or to support a 510(k) submission. The study will be conducted at one site: Stanford University.

This study will enroll 24 subjects (as per FDA approval) to establish the maximum length of Lantern infusion set wear when 80% of sets are still functional (excluding accidental "pull-outs"). Each participant will place the set and wear it for 10 days or until set failure and data will be collected on the cause of set failure. If a set is accidentally pulled out, it can be replaced by the subject. Failures are based on:

1. Presence of serum ketones with hyperglycemia
2. Unexplained hyperglycemia
3. Signs of infection at the infusion site
4. Pump occlusion alarm
5. Adhesive failure

Since infusion set failures will occur after variable lengths of wear, regularly scheduled visits are unlikely to capture the day of an infusion set failure. Instead the subject will be taught how to insert the set, measure erythema and induration with a ruler marked in millimeters and to take a picture of the infusion site. Subjects will be instructed to text the study team when they remove their infusion set and to send a picture of the infusion site and measurements. If there is any evidence of an infection (≥10 mm of erythema or induration), they will be asked to come in that day for an unscheduled visit.

ELIGIBILITY:
Inclusion Criteria:

Type 1 Diabetes by clinical definition

1. Age 22 and over
2. On tethered insulin pump therapy for at least 3 months using Lispro or Aspart insulin.
3. Hemoglobin A1c level less than or equal to 9%
4. Eating more than 60 grams of carbohydrate each day
5. For females, not currently known to be pregnant
6. Understanding and willingness to follow the protocol and sign informed consent
7. Willingness to wear the experimental infusion sets
8. Willingness to have photographs taken of their infusion sites
9. Ability to speak, read and write in the language of the investigators

Exclusion Criteria:

The presence of any of the following is an exclusion for the study:

1. Diabetic ketoacidosis in the past 3 months
2. Severe hypoglycemia resulting in seizure or loss of consciousness within 3 months prior to enrollment
3. Pregnant or lactating
4. Known tape allergies
5. Active infection
6. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol
7. Known cardiovascular events in the last 6 months
8. Known acute proliferative diabetic retinopathy
9. Known adrenal disorder
10. Current treatment for a seizure disorder
11. Inpatient psychiatric treatment in the past 6 months
12. Lack of stability on medication 1 month prior to enrollment including antihypertensive, thyroid, anti-depressant or lipid lowering medication.
13. Use of SGLT inhibitor
14. Suspected drug or alcohol abuse
15. Dialysis or end stage kidney disease

Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Buckingham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lal RA, Hsu L, Zhang J, Schondorff PK, Heschel M, Buckingham B. Longevity of the novel ConvaTec infusion set with Lantern technology. Diabetes Obes Metab. 2021 Aug;23(8):1973-1977. doi: 10.1111/dom.14395. Epub 2021 Apr 18. PMID 33822472

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lantern Infusion Set
Started | 24
Completed | 22
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis for baseline characteristics.
Arm/Group | Lantern Infusion Set
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Diabetes Duration [Mean (Standard Deviation); unit: years] | 26.4 (12.2)
HbA1c [Mean (Standard Deviation); unit: % glcosylated HBG:total HBG] | 7.1 (0.8)
Total Daily Insulin Dose (Units) [Mean (Standard Deviation); unit: units] | 48.0 (16.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Time to Infusion Set Failure
Description: Time to when the infusion set fails and needs to be replaced.
Time Frame: 10 days of infusion set wear
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lantern Infusion Set
Number analyzed (Participants) | 22
days | 8.0 (2.4)

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Lantern Infusion Set
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 12/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lantern Infusion Set (N=24)
subcutaneous infection (Skin and subcutaneous tissue disorders) | 1 (1)
hyperglycemia (Endocrine disorders) | 6 (6) — hyperglycemia unresponsive to a correction dose of insulin
ketotosis (Endocrine disorders) | 1 (1) — ketosis with hyperglycemia
adhesive failure (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03819634/Prot_SAP_000.pdf